CLINICAL TRIAL: NCT05927402
Title: Effect of Laughter Therapy Based on Kolcaba Comfort Theory on Surgical Stress, Oxygen Saturation, Pain and Comfort Level in Bariatric Surgery Patients
Brief Title: Effect of Laughter Therapy on Surgical Stress, Oxygen Saturation, Pain and Comfort Level
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Gülşah Kayserilioğlu, Lecturer, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ANKARAYBU-GKAYSERILIOGLU-001
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Bariatric Surgery Pateints; Lauhgter Therapy; Laughter Yoga
Keywords: bariatric surgery patients; laughter therapy; laughter yoga

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Laughter Therapy Based on Kolcaba Comfort Theory — The laughter yoga will be applied to experimanetal group. Every laughter yoga practice is 45 minutes long and is planned 3 times a week for a total of 6 sessions. Control group patients will take only routine nursing care.

SUMMARY:
The aim of this study is to examine the effect of laughter therapy based on Kolcaba comfort theory, on surgical stress, oxygen saturation, pain and comfort level in bariatric surgery patients. The main questions it aims to answer are:

1. Is there a significant difference between salivary cortisol levels of patients with and without laughter yoga before surgical intervention?
2. Is there a significant difference between the blood glucose levels of patients who were and were not treated with laughter yoga before surgical intervention?
3. Is there a significant difference between the mean scores on the perceived stress scale of patients who were and were not treated with laughter yoga before surgical intervention?
4. Is there a significant difference between the oxygen saturation levels of patients with and without laughter yoga before surgical intervention?
5. Is there a significant difference between the mean scores on the comfort level scale of patients who were and were not treated with laughter yoga before surgical intervention?
6. Is there a significant difference between the mean scores on the pain scale of patients who were and were not treated with laughter yoga before surgical intervention?

The study population will consist of patients who will apply to the general surgery clinic of Düzce University Research and Application Center between June 2023 and April 2024, who will undergo bariatric surgery and agree to participate in the study. The data collected from these patients will be analyzed.

From the patients who meet the inclusion criteria and agree to participate in the study; experimental and control groups will be determined by simple randomization. They will be informed about the research (a 15-minute presentation prepared by the researcher explaining what laughter therapy is) and their verbal and written permission will be obtained.

The laughter yoga will be applied to experimanetal group. Every laughter yoga practice is 45 minutes long and is planned 3 times a week for a total of 6 sessions. Control group patients will take only routine nursing care.

ELIGIBILITY:
Inclusion Criteria:

* Those who can speak and understand Turkish,
* Those who agreed to participate in the study,
* Adult age group between 18 and 60 years old,
* Those with pain intensity <2 according to the Visual Comparison Scale,
* Those with time and place orientation,
* Those without vision and hearing problems,
* Those who are literate or have literate relatives,
* Those without history of psychiatric illness,
* Those without any history of psychotropic drug use and history,
* Those without previous laughter yoga practice,
* Those with a smartphone/computer/tablet,
* Those who undergone laparoscopic sleeve gastrectomy surgery,
* Those who can attend the trainings at the specified times so that cortisol is not affected by circadian rhythm,
* Those who are able to comply with the collection of saliva samples,
* American Society of Anesthesiologist (ASA) score I, II or III as assessed by physicians

Exclusion Criteria:

* Those who speak Turkish but cannot understand,
* Those who are under 18 and over 60 years of age,
* Those who are not willing to participate in the study,
* Those diagnosed with psychiatric illness,
* Those with previous laughter yoga practice,
* Those with physical limitations/respiratory problems who cannot perform yoga movements,
* Those who have difficulty in doing breathing exercises due to deviated septum etc,
* Those who have undergone abdominal surgery in the last six months
* Hypothyroidism, hyperaldosteronism, pregnancy, malignancy, congestive heart failure, psychotic disorder, chronic liver failure, uncontrolled hypertension, glaucoma, herniation, nephrotic syndrome, type 2 diabetes mellitus, Patients with a diagnosis of chronic renal failure and continuous use of medication were excluded as salivary cortisol levels may be affected,
* Those with an ASA score of 4,
* Those who don't undergone laparoscopic sleeve gastrectomy surgery,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-07-03 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Stress level | before first laughter therapy application
  with Perceived Stress Scale-14, 0-56 (min-max), higher scores mean worse outcome
Stress level | after sixth laughter therapy application (preop first day)
  with Perceived Stress Scale-14, 0-56 (min-max), higher scores mean worse outcome
Stress level | postop first day
  with Perceived Stress Scale-14, 0-56 (min-max), higher scores mean worse outcome
Pain level | before first laughter therapy application
  with Visual Analog Scale, 0-10 (min-max), higher scores mean worse outcome
Pain level | after sixth laughter therapy application (preop first day)
  with Visual Analog Scale, 0-10 (min-max), higher scores mean worse outcome
Pain level | postop first day
  with Visual Analog Scale, 0-10 (min-max), higher scores mean worse outcome
Comfort level | before first laughter therapy application
  with General Comfort Questionaire, 48-192 (min-max), higher scores mean worse outcome
Comfort level | after sixth laughter therapy application (preop first day)
  with General Comfort Questionaire, 48-192 (min-max), higher scores mean worse outcome
Comfort level | postop first day
  with General Comfort Questionaire, 48-192 (min-max), higher scores mean worse outcome
Blood glucose level | before first laughter therapy application
  with blood glucose meter
Blood glucose level | after sixth laughter therapy application (preop first day)
  with blood glucose meter
Blood glucose level | postop first day
  with blood glucose meter
Oxygen Saturation Level | before first laughter therapy application
  with pulse oximetry
oxygen saturation level | after sixth laughter therapy application (preop first day)
  with pulse oximetry
Oxygen Saturation Level | postop first day
  with pulse oximetry
salivary cortisol sample | before first laughter therapy application
  salivette cortisol
salivary cortisol sample | after sixth laughter therapy application (preop first day)
  salivette cortisol
salivary cortisol sample | postop first day
  salivette cortisol

CONTACTS AND LOCATIONS:
Locations (1):
- Düzce University Research and Application Center, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No